CLINICAL TRIAL: NCT06890182
Title: Firmonertinib Combine With Carboplatin/Cisplatin and Pemetrexed as Neoadjuvant Therapy for Resectable Stage Ⅱ-ⅢB EGFR Sensitive Mutanted NSCLC
Brief Title: Firmonertinib Combined With Chemotherapy as Neoadjuvant Therapy for Resectable Stage Ⅱ-ⅢB EGFR Sensitive Mutanted NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20250016
Record Dates: First submitted 2025-03-16; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Firmonertinib combined with Carboplatin/Cisplatin and Pemetrexed (Experimental): furmonertinib 80mg/d for 12 weeks and carboplatin AUC5 d1 iv / cisplatin 75mg/m2 d1 iv+ pemetrexed 500mg/m2 d1 iv at 21 day cycles for 4 cycles
  Interventions: Drug: Firmonertinib combined with Carboplatin/Cisplatin and Pemetrexed

INTERVENTIONS:
Drug: Firmonertinib combined with Carboplatin/Cisplatin and Pemetrexed — furmonertinib 80mg/d for 12 weeks and carboplatin AUC5 d1 iv / cisplatin 75mg/m2 d1 iv+ pemetrexed 500mg/m2 d1 iv at 21 day cycles for 4 cycles

SUMMARY:
This is a phase II study aimed to assess the efficacy and safety of firmonertinib combined with carboplatin/cisplatin and pemetrexed as neoadjuvant therapy in stage II-IIIB resectable NSCLC patients.

DETAILED DESCRIPTION:
In this open-label, single-arm, phase 2 study, 31 eligible patients with EGFR mutated stage IIIA-IIIB resectable NSCLC will be recruited to receive firmonertinib for 12 weeks combined with carboplatin/cisplatin and pemetrexed for 4 cycles (21 d/cycle) as neoadjuvant therapy before radical surgery. Radiological and pathological evaluations will be performed before and after the neoadjuvant therapy to assess the efficacy of treatment. Adverse events during neoadjuvant therapy, disease and survival status will also be collected in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed consent prior to any study specific procedures
2. at least 18 years of age
3. Histology or cytology diagnose of non-small cell lung cancer within 60 days
4. ECOG PS of 0 to 1 at screening with no clinically significant deterioration in the previous 2 weeks
5. Stage II-IIIB NSCLC that is expected to be resectable, as assessed by the investigator (8 thUICCTNM staging),
6. According to RECIST 1.1, patients have at least one measureable tumor lesion (The longest axis ≥10mm)
7. EGFR mutation positive (exon 19 deletions or exon 21 L858R, with or without other EGFR mutations)
8. Without prior anti-tumor treatment
9. Withe adequate organ function of hematology, liver and kidney
10. Using adequate and effective contraception, Male patients should be use condoms; women should refrain from breastfeeding and have a negative pregnancy test prior to the first administration of the study drug if within during child-bearing age

Exclusion Criteria:

1. Dual or multiple primary NSCLC
2. Any prior anti-tumor treatment
3. With history of other malignancy except for radical resected tumors without recurrence for 5 years or more
4. Diseases or clinical states with severe abnormalities of gastrointestinal function that may interfere with the ingestion, transit, or absorption of the study drug.e.g., inability to take medication orally, uncontrolled nausea and vomiting
5. With severe or uncontrolled systemic disease such as uncontrolled hypertention, diabetes mellitus, chronic heart failure, unstable angina, myocardial infarction within 1 year, active hemorrhage, active HBV/HCV/HIV or other infections requiring infusion treatment
6. Laboratory tests indicate insufficient bone marrow reserve or organ reserve
7. Women with pregnancy or breastfeeding
8. Patients with known or suspected drug allergies, or other contraindications
9. Other conditions that, in the opinion of the investigator, make participation in this trial inappropriate
10. Patients who are currently or previously enrolled in any other anti-tumor clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Major pathological response rate (MPR) | Approximately 24 weeks following the first dose of study drug
  Proportion of resected specimens with ≤10% residual tumor cells assessed by surgical specimen pathology

SECONDARY OUTCOMES:
Pathological Complete Response Rate（pCR) | Approximately 24 weeks following the first dose of study drug
  The proportion of patients with pathological response rate in the resected tumor.
Objective Response Rate (ORR) | Approximately 8 weeks following the first dose of study drug
  According to RECIST 1.1 criteria, after 8 weeks of neoadjuvant therapy CT scans scans assessed the proportion of patients in partial and complete remission.
Rate of R0 Resection | Approximately 16 weeks following the first dose of study drug
  The proportion of patients with R0 resection.
Pathological downstaging of lymph node rate | Approximately 16 weeks following the first dose of study drug
  The proportion of patients with pathological downstaging of lymph node rate
Incidence of adverse events (AE) | Approximately 12 weeks following the first dose of study drug
  The number of patients with adverse events and the severity according to CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Zhansheng Jiang, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital